CLINICAL TRIAL: NCT06242522
Title: Fertility and Pregnancy After Avelumab Treatment
Acronym: FERTILAVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL24_0089
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Gestational Trophoblastic Tumours; Immune Checkpoint Inhibitors
Keywords: Immune checkpoint inhibitors; Gestational trophoblastic tumours; Young women; Childbearing age; Pregnancy
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Intervention Model Description: Prospective and retrospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female patients with gestational trophoblastic tumour. (Other): Female patients treated in phase II or III clinical trials: TROPHIMMUN and TROPHAMET or who have received AVELUMAB outside the trial for a gestational trophoblastic tumour.
  Interventions: Other: Telephone interview

INTERVENTIONS:
Other: Telephone interview — Collection of gynaecology-obstetrics data on patients treated with AVELUMAB

SUMMARY:
Immune checkpoint inhibitors (ICIs), such as anti-PD-1/PD-L1 agents, initially evaluated in advanced non-curative pathologies, are now being evaluated in adjuvant or even neoadjuvant curative treatment conditions. This paradigm shift is leading to the treatment of young women, particularly in the context of gestational trophoblastic tumours. Given the potential autoimmune side-effects affecting endocrine functions, as well as their impact on maternal-foetal tolerance mechanisms, accurate assessment of post-ICT fertility is necessary. In the coming years, treatment with anti-PD-L1 (avelumab) could become a cornerstone of the therapeutic strategy for patients with gestational trophoblastic tumours.

However, these patients are often young and of childbearing age, so safety of use in terms of fertility and successful pregnancies is an essential factor in the widespread use of immunotherapy as a treatment option. Some studies have reported the possibility of conceiving after avelumab treatment, but no cohort has been reported. This study aims to explore fertility and the course of potential pregnancy in 50 patients treated with anti-PD-L1 (avelumab) over the last 5 years in several French centres.

ELIGIBILITY:
* Inclusion Criteria :

  * Patient aged over 18 years
  * Have received AVELUMAB treatment for GTT in the TROPHIMMUN or TROPHAMET trials, or have received AVELUMAB outside the trial for gestational trophoblastic tumour.
  * Did not object to participating in the study
* Exclusion Criteria :

  * Patient who has died
  * Patient who has had a hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Describe the time to pregnancy in patients treated with anti PDL1 (avelumab) for GTT | Up to 5 years
  Time to achieve pregnancy after stopping contraception

CONTACTS AND LOCATIONS:
Locations (1):
- Centre De Reference Des Maladies Trophoblastiques, Hôpital Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No